CLINICAL TRIAL: NCT04124978
Title: Evaluation of the Effectiveness of Direct to Consumer Mandibular Advancement Devices as an Adjunct for the Treatment of Mild to Moderate Obstructive Sleep Apnoea (OSA)
Brief Title: Evaluation of Prefabricated Adjustable Thermoplastic Mandibular Advancement Devices for Obstructive Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/3100
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; mandibular advancement device; thermoplastic; adjustable; MyTAP
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention group (Experimental): prospective, single armed, single centre trial study using the MyTAP device on a daily basis for a period of 3 months
  Interventions: Device: mandibular advancement device

INTERVENTIONS:
Device: mandibular advancement device — use of prefabricated adjustable mandibular advancement device to improve OSA

SUMMARY:
Use of mandibular advancement devices(MADs) in the treatment of Obstructive Sleep Apnea is established, however this is hampered by high costs, long wait times and non-assured success in the local Asian setting. There are few studies which look at the use of prefabricated thermoplastic mandibular devices with a titratable component and its efficacy. In addition, it is direct-to-consumer and an economical option, thus there may be a role in the use of such devices to better select patients who may benefit and are thinking of using MADs.

The investigators aim to evaluate the effectiveness of the use of Prefabricated adjustable thermoplastic mandibular advancement devices(PAT-MADs)(MyTAP) in the treatment of OSA and its role for predicting treatment success in an Asian population.

DETAILED DESCRIPTION:
Mandibular advancement devices (MAD) serve as an adjunct to the treatment of snoring as well as mild-moderate OSA. It is widely accepted that upper airway muscle activity decreases during sleep, leading to increased collapsibility of the pharyngeal tissues, mandibular opening and posterior displacement of the tongue. These changes result in narrowing of the oropharyngeal and hypopharyngeal airway (Hudgel 1992). Their primary action is to advance the mandible and tongue to increase the upper airway size. Recent systemic review on the effectiveness of MAD in treating OSA by Torres et al in the Laryngoscope showed that 16 out of 18 large scale studies showed significant improvement in Apnea-Hypopnea index (AHI).

There are a wide variety of MAD commercially available and they can be broadly divided into custom made vs prefabricated makes as well as titratable versus non-titratable types. It is shown that custom made, titratable fitted MADs are superior in efficacy as compared to their counterpart models. However, high cost, delayed waiting times and multiple clinic visits are required for patients to be fitted with custom MADs by a professional orthodontist. Newly developed direct to consumer thermoplastic MADs (MyTap) brings the benefit of mouldable bite and form "custom" fit with the option of titration to the user at a lower cost, technical ease of use and fit in the clinic setting.

Participants who are diagnosed with simple snoring or mild to moderate OSA are able to trial use thermoplastic MADs to have a sense of the level of comfort and effectiveness MAD can bring to improve their OSA, serving as a bridging device prior to committing to the use of custom made MAD.

The investigators aim to evaluate the effectiveness of the use of Prefabricated adjustable thermoplastic mandibular advancement devices(PAT-MADs)(MyTAP) in the treatment of OSA and its role for predicting treatment success, compliance and comfort in an Asian population.

ELIGIBILITY:
Inclusion Criteria:

* 18years old and above
* English competency
* Formal diagnosis of mild-moderate OSA on PSG
* Ability to provide informed consent

Exclusion Criteria:

* diagnosed severe OSA
* evidence of central sleep apnea events
* dental conditions which preclude proper use of the MAD
* treatment with other devices (e.g. tongue retainers, PAP therapy)
* pregnancy
* known allergic reactions to the components of the study product were excluded from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 3 months
  apnea-hypopnea index
Apnea index (AI) | 3 months
  apnea index
Hypopnea index (HI) | 3 months
  Hypopnea index
Oxygen disturbance index (ODI) | 3 months
  Oxygen disturbance index
Lowest oxygen saturation (Lsat) | 3 months
  Lowest oxygen saturation
Epworth sleepiness score (ESS) | 3 months
  Epworth sleepiness score measures the level of sleepiness in a participant. Minimum value of 0 to a maximum level of 24, whereby the higher the value, the sleepier the participant.
Abbreviated functional outcomes of sleep questionnaire (FOSQ-10) | 3 months
  Quality of life survey made of up 10 self rated questions which assess the quality of sleep in participants with sleep disorders. Minimum value is 0 and maximum value is 40, where the lower the global value, the worse off the quality of sleep.
Pittsburgh sleep quality index (PSQI) | 3 months
  Quality of life survey made up of 19 self rated questions which assesses the quality of 7 different aspects of sleep in participants with sleep disorders. Minimum value is 0 and maximum value is 21, where the higher the global value, the more severe the difficulties in different aspects of sleep.

SECONDARY OUTCOMES:
Predicting future use | 3 months
  if the use of PAT-MAD is an acceptable treatment to patients who are keen to try customizable MAD but are unsure of the treatment suitability and effectiveness for their OSA, in the form of adherence, self/3rd party reported symptom improvement and ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Toh Song Tar, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soh L, Han HJ, Yue Y, Tay JY, Hao Y, Toh ST. Evaluation of prefabricated adjustable thermoplastic mandibular advancement devices (PAT-MADs) for obstructive sleep apnea: an Asian experience. Sleep Med. 2020 Nov;75:96-102. doi: 10.1016/j.sleep.2020.02.025. Epub 2020 Mar 7. PMID 32853924